CLINICAL TRIAL: NCT05498753
Title: Development, ADL, Participation, and Quality of Life in Preterm Infants: A Longitudinal Follow Up Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202101737B0
Record Dates: First submitted 2022-02-17; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-02

CONDITIONS: Preterm Birth
Keywords: Body function and body structure; Participation; Life activities; Quality of Life
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Healthy infants
- Experimental: Preterm Infants

SUMMARY:
A Longitudinal Study of Function, ADL, and Quality of life of Patients with Developmental Disabilities

DETAILED DESCRIPTION:
Preterm Infant is defined as a group of patients whose gestational age is lower than 37 weeks due to either iatrogenic reasons or maternal reasons. Preterm infant could be classified into 4 group according to gestational age: very early preterm infant, early preterm infant, midterm preterm infant, and late preterm infant. Moreover, they could be categorized into 3 groups of birth weight: extremely low birth weight, very low birth weight, and low birth weight. These varies of preterm infant are indicated to have further developmental and body-functional difficulties and lags. Under the basis of International Classification of Functioning, Disability and Health-Children and Youth Version (ICF-CY) framework, problems related to Preterm infant would further limit their activities of daily living (ADL), participation, and health related quality of life (HRQOL).

The three fundamental goals of early rehabilitation for preterm infant after leaving NICU are: optimizing function within each child's prognostic potential, preventing the development of secondary conditions that impact life-long health, and promoting children's participation and qualities in their lives. Understanding knowledges of these developmental patterns of Function and Participation in Life Activities (FPLA) and HRQOL may be helpful for anticipating and managing the problems. This study hypothesizes that the course of developmental patterns in FPLA and HRQOL of preterm infant evolve with their age. The functional recovery levels include developmental function, activity, participation, and quality of life (QOL).

This study included validity and reliability study and a prospective 2 phases, 3-years period longitudinal study of patient with preterm infant. From the first half year, 50 used-to-be preterm infant children and 50 used-to-be full-term infant children will be recruited to examine the reliability and validity of assessment tools and examiner. From the late half of the 1st and following years, 100 used-to-be full-term infant children (0-3 years old) and 200 used-to-be preterm infant children will be recruited for follow up research. All participants will receive a series of FPLA and HRQOL assessments, which are based on ICF-CY framework. Examiners will select assessment tools that appropriate to participant's age. Moreover, during this prospective longitudinal study, each participant will receive FPLA and HRQOL assessments as baseline, and re-evaluation every 6-months after the first data collection point. We believe the results of this study will refine services and supports for children with preterm infant to meet these goals.

ELIGIBILITY:
Inclusion Criteria:

* Children who were born before 37 weeks
* Age 0-3 y/o
* Agree to sign inform consent

Exclusion Criteria:

* Active medical condition (e.g. infection)
* Concurrent disease which affect nuerological development, such as cerebral palsy, or other disease not typically associated with preterm

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Enroll preterm and healthy infants.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-02-21 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline general development for Healthy child and preterm infants at 6 months 1 | From 6 months to 4 years
  Bayley scales of infant and Toddler Developmentfourth edition is used to examine the body function, motor function, cognitive, language, and social behavior.
  (Scores from 0 to 140, higher scores mean a better outcome.)
Change from baseline general development for Healthy child and preterm infants at 6 months 2 | From 6 months to 4 years
  Comprehensive Development Inventory for Infant and Toddlers (CDIIT) is used to examine the body function, motor function, cognitive, language, and social behavior.
  (Higher scores mean a better outcome.)
Change from baseline general development for Healthy child and preterm infants at 6 months 3 | From 6 months to 4 years
  Hawaii Early Learning Profile (HELP) is used to examine the regulatory/sensory orginization, motor function, cognitive, language, and social behavior, and self-help. (Higher scores mean a better outcome.)
Change from baseline general development for Healthy child and preterm infants at 6 months 4 | From 6 months to 4 years
  General Movements Assessment (GMA) is used to examine the motor function. (Higher scores mean a better outcome.)
Change from baseline functions for preterm infants at 6 months | From 6 months to 4 years
  PREMature Infant Index(PREMII) is used to examine the respiratory support, oxygen administration, apnea, bradycardia, desaturation, thermoregulation, feeding, and weight.
  (Higher scores mean a better outcome.)

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ling Chen, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No